CLINICAL TRIAL: NCT05405036
Title: The Psychometric Properties of the Turkish Version of Interpersonal Communication Questionnaire in Physiotherapy Students
Brief Title: The Psychometric Properties of the Turkish Version of Interpersonal Communication Questionnaire
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Other Study IDs: ATADEK-2022/08/01
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Educational Problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students: 60 second-year students studying at the Department of Physiotherapy and Rehabilitation at University are planned to attend.
  Interventions: Other: simulated patient

INTERVENTIONS:
Other: simulated patient — In the last month of the Measurement and Evaluation course in Physiotherapy, a simulated patient session will be held four times (with disease in the cervical-lumbar-shoulder and knee region). Students will be evaluated by the methods they learned about patients. 10 days before and after the simulated patient sessions, the questionnaire will be applied in Turkish for validity and reliability, and then the questionnaire will be repeated after the simulated patient sessions are over, and the effect of the smile patient sessions on the perceived communication skills of the patient will be examined.

SUMMARY:
In a study conducted by Lewis et al. in 2008, an "interpersonal communication" questionnaire was developed to measure the perceived interpersonal skills of physiotherapy and rehabilitation students regarding patient interaction. It was determined that the questionnaire used especially after the simulated patient training increased the communication of physiotherapy and rehabilitation students after the simulated patient training. However, the questionnaire was not translated into Turkish and its validity and reliability were not investigated. Therefore, in this study, the authors aim to investigate the Turkish validity and reliability of the Interpersonal Communication Questionnaire as the primary purpose. Secondly, to investigate the effect of simulated patient experience on the perceived interpersonal skills of physiotherapy and rehabilitation students regarding patient interaction at the time of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Students taking the Measurement and Evaluation II course in Physiotherapy and Rehabilitation

Exclusion Criteria:

* Not volunteering
* Those who are being treated with any psychiatric diagnosis
* Students who fail the course or fail to pass it successfully

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 second year students aged 18-23 studying at the physiotherapy and rehabilitation department of Acibadem mehmet ali aydınlar university are planned to participate in the research.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Interpersonal Communication Questionnaire | Change from Baseline Scores at 2 week and 6. week
  Eight statements were constructed; four related to a sub-scale measuring factors associated with communication anxiety, and four related to communication confidence.
  Each statement had a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree. Sub-scale scores ranged from a possible 4-20; a higher score indicating either higher levels of communication confidence or anxiety.

SECONDARY OUTCOMES:
Visual Analog Scale | Change from Baseline Scores at 6. week
  A visual analog scale between 0 and 10 will be used to evaluate communication anxiety, stress, motivation and success that may occur when students go into clinical practice at the beginning and end of the term and when they meet with the patient.Zero will be determined to be none at all, and 10 to the maximum I can think of
Interpersonal Communication Competence Inventory | Change from Baseline Scores at 6. week
  Huang and Lin (18) developed the CITI based on four basic skill areas (listening skill, empathy skill, expression skill, social relaxation skill) in order to evaluate the communication competence of university students in accordance with the relational approach.The scores that can be obtained from the measurement tool vary between 15 and 75. Items 10 and 13 are reverse scored. A high score on the measurement tool indicates a high level of interpersonal communication competence.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ALACA, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided